CLINICAL TRIAL: NCT00224016
Title: A Multi-Center, Open-Label (OL), Active-Controlled, Dose-Titration Study Evaluating the Safety, Efficacy and PK of Oxybutynin Transdermal Systems in the Treatment of Detrusor Overactivity in Pediatric Patients
Brief Title: Safety and Efficacy Study of Transdermal Oxybutynin to Treat Overactive Bladder With a Neurological Condition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O03010
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Detrusor Hyperreflexia
MeSH Terms: interventions — oxybutynin; Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxybutynin Transdermal System (Experimental): Oxybutynin Transdermal System 1.3 mg/day, 2.6 mg/day, or 3.9 mg/day
  Interventions: Drug: Oxybutynin
- Oral oxybutynin (Active Comparator): 5 to 15 mg/day immediate release or extended release tablets, or syrup
  Interventions: Drug: Oxybutynin

INTERVENTIONS:
Drug: Oxybutynin — 1.3, 2.6, 3.9 mg/day transdermal
  Other Names: Oxytrol
  Arms: Oxybutynin Transdermal System
Drug: Oxybutynin — 5 to 15 mg/day immediate release or extended release tablets, or syrup
  Other Names: Ditropan, Ditropan XL, Oxybutynin
  Arms: Oral oxybutynin

SUMMARY:
This study will evaluate the safety and effectiveness of an anticholinergic drug treatment administered by transdermal patch to treat overactive bladder in children who have a neurological condition (e.g. spina bifida) that contributes to their overactive bladder.

DETAILED DESCRIPTION:
This study will use a multicenter, randomized, open-label, active-controlled, dose-titration, parallel group design, in approximately pediatric patients with detrusor overactivity associated with a neurological condition.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient with a diagnosis of detrusor overactivity associated with a neurological condition;
* Use clean intermittent catheterization
* On stable dose of oral oxybutynin before participation

Exclusion Criteria:

* Have one or more treatable conditions, other than neurogenic bladder dysfunction, that may cause urinary incontinence or urgency
* Have any medical condition that precludes their participation in the study or may confound the outcome of the study

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2004-12; Primary Completion 2007-04 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hoel, RPh, PhD, Study Chair — Watson Laboratories, Inc.
Locations (23):
- United States (23):
  - Watson Investigational Site, Little Rock, Arkansas
  - Watson Investigational Site, Orange County, California
  - Watson Investigational Site, San Diego, California
  - Watson Investigational Site, Denver, Colorado
  - Watson Investigational Site, Washington D.C., District of Columbia
  - Watson Investigational Site, Detroit, Michigan
  - Watson Investigational Site, Minneapolis, Minnesota
  - Watson Investigational Site, Jackson, Mississippi
  - Watson Investigational Site, Kansas City, Missouri
  - Watson Investigational Site, St Louis, Missouri
  - Watson Investigational Site, Voorhees Township, New Jersey
  - Watson Investigational Site, Albany, New York
  - Watson Investigational Site, Buffalo, New York
  - Watson Investigational Site, Poughkeepsie, New York
  - Watson Investigational Site, Ashville, North Carolina
  - Watson Investigational Site, Durham, North Carolina
  - Watson Investigational Site, Columbus, Ohio
  - Watson Investigational Site, Oklahoma City, Oklahoma
  - Watson Investigational Site, Hershy, Pennsylvania
  - Watson Investigational Site, Dallas, Texas
  - Watson Investigational Site, Houston, Texas
  - Watson Investigational Site, Plano, Texas
  - Watson Investigational Site, Salt Lake City, Utah

REFERENCES:
- [Result] Cartwright PC, Coplen DE, Kogan BA, Volinn W, Finan E, Hoel G. Efficacy and safety of transdermal and oral oxybutynin in children with neurogenic detrusor overactivity. J Urol. 2009 Oct;182(4):1548-54. doi: 10.1016/j.juro.2009.06.058. Epub 2009 Aug 15. PMID 19683731

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxybutynin TDS: Oxybutynin Transdermal System
- Oral Oxybutynin: Oxybutynin tablets
Period: Titration Period
Arm/Group | Oxybutynin TDS | Oral Oxybutynin
Started | 39 | 16
Completed | 38 | 15
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Maintenance Period
Arm/Group | Oxybutynin TDS | Oral Oxybutynin
Started | 38 | 15
Completed | 36 | 14
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Follow-Up Period
Arm/Group | Oxybutynin TDS | Oral Oxybutynin
Started | 35 | 0 (This group of subjects did not proceed to follow-up period.)
Completed | 35 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxybutynin TDS | Oral Oxybutynin | Total
Number analyzed (Participants) | 39 | 16 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 16 | 55
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.2 (2.64) | 11.8 (2.82) | 10.6 (2.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 22 | 5 | 27
Region of Enrollment [Number; unit: participants]
  United States | 39 | 16 | 55

OUTCOME MEASURES:

1. Primary Outcome: Average Catheterization Urine Volume
Description: Change from baseline in average volume of urine collected by catheterization
Time Frame: 14 weeks
Population: Modified intent-to-treat (mITT) population, Last Observation Carried Forward (LOCF) imputation
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Oxybutynin TDS | Oral Oxybutynin
Number analyzed (Participants) | 38 | 14
mL
  Baseline Catheterization Volume | 95.3 (63.88) | 114.0 (74.67)
  Change from Baseline in Cath Volume | 30.0 (46.20) | 52.4 (50.45)

2. Secondary Outcome: Catheterizations Without Leakage
Description: Percentage of catherizations without leakage
Time Frame: 14 weeks
Population: mITT, LOCF
Measure: Mean (Standard Deviation); unit: % of participants
Arm/Group | Oxybutynin TDS | Oral Oxybutynin
Number analyzed (Participants) | 38 | 14
% of participants
  Baseline % Catheterizations without leakage | 28.7 (34.85) | 38.1 (41.86)
  Endpoint % Catheterizations without leakage | 53.8 (36.05) | 72.6 (26.44)

3. Secondary Outcome: Urine Volume After First Awakening
Description: Change from baseline in average volume of urine collected after first morning awakening
Time Frame: 14 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: mL

ADVERSE EVENTS:
Arm/Group | Oxybutynin TDS | Oral Oxybutynin
Serious Adverse Events (participants affected / at risk) | 6/39 | 3/16
Other Adverse Events (participants affected / at risk) | 33/39 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin TDS (N=39) | Oral Oxybutynin (N=16)
Allergic reaction (General disorders) | 0 (0) | 1 (1)
Knee wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Worsening abdominal pain (General disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Cardiac disorders) | 0 (0) | 1 (1)
VP shunt malfunction (Nervous system disorders) | 2 (2) | 1 (1)
Worsening dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tethered cord (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin TDS (N=39) | Oral Oxybutynin (N=16)
Fever (General disorders) | 6 (7) | 3 (4)
Headache (General disorders) | 7 (12) | 2 (3)
Urinary tract infection (Infections and infestations) | 6 (6) | 2 (2)
Infection (Infections and infestations) | 7 (8) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pain abdominal (General disorders) | 3 (3) | 2 (2)
Pain back (General disorders) | 3 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 4 (7) | 2 (3)

LIMITATIONS AND CAVEATS:
The transdermal groups included more males and younger subjects. The study was not designed to compare the transdermal and oral groups. Advserse event data reported for the titration and maintenance periods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less